CLINICAL TRIAL: NCT00089700
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Three-Arm Study of the Anti-CD4 Monoclonal Antibody TNX-355 With Optimized Background Therapy in Treatment-Experienced Subjects Infected With HIV-1
Brief Title: TNX-355 With Optimized Background Therapy (OBT) in Treatment-Experienced Subjects With HIV-1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tanox (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TNX-355.03
Record Dates: First submitted 2004-08-10; First posted 2004-08-12 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-02

CONDITIONS: HIV Infections
Keywords: HIV; AIDS; Treatment Experienced; Optimized Background Therapy; HIV-1
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — ibalizumab

INTERVENTIONS:
Drug: TNX-355

SUMMARY:
This is a 48-week study to compare TNX-355 plus OBT to placebo plus OBT in HIV subjects. You must have a stable viral load of at least 10,000 copies/ml, been treated with highly active antiretroviral therapy (HAART) for at least 6 months, be triple class experienced, and presently failing or have failed a HAART regimen. Subjects will receive infusions every week for 8 weeks, then every two weeks.

DETAILED DESCRIPTION:
This 48-week, multicenter, randomized, double-blinded, placebo-controlled, multi-dose, three-arm safety and efficacy study of approximately 80 subjects will compare TNX-355 plus OBT to placebo plus OBT in adult subjects infected with HIV-1. Subjects must: 1) have a stable viral load of 10,000 copies/mL, determined within 8 weeks prior to randomization (Day 1); 2) have been treated with HAART for at least 6 months (cumulatively); 3) be triple class experienced, with historical evidence of exposure to each of the three traditional classes of antiretroviral therapy (ART): nucleoside reverse transcriptase inhibitors (NRTIs), non-nucleoside reverse transcriptase inhibitors (NNRTIs), and protease inhibitors (PIs); and 4) be presently failing or have failed a HAART regimen within 8 weeks prior to screening (Screening visit 1).

Subjects will be assigned to OBT based upon their past medication history and the results of the virus sensitivity testing (PSGT, ViroLogic, Inc.), and then randomized to a study arm to begin receiving OBT plus study medication at the Day 1 visit. Fusion/entry inhibitors will not be permitted as part of the optimized background therapy. All subjects will be randomized equally (1:1:1 ratio), in a double-blinded fashion, among three arms to receive OBT plus one of the following: Arm A, alternating intravenous infusions of TNX-355, 15 mg/kg and placebo weekly for the first 9 doses (through the Week 8 visit), and then intravenous infusions of TNX-355, 15 mg/kg every two weeks; Arm B, TNX-355, 10 mg/kg intravenous infusions weekly for the first 9 doses (through the Week 8 visit), and then intravenous infusions of TNX-355, 10 mg/kg every two weeks; or Arm C, weekly intravenous infusions of placebo for the first 9 doses (through the Week 8 visit), and then intravenous infusions of placebo every two weeks.

Subjects will continue to receive blinded therapy until that therapy fails. Subjects that do not achieve a viral load reduction of at least 0.5 log10 from their baseline value on two consecutive protocol-defined assessments after Week 12 will be considered virologic failures. Subjects that experience virologic failure after Week 16 (i.e., earliest point at which virologic failure can be confirmed after Week 12) will have the option of being assigned to new OBT plus open-label TNX-355 given as a 15 mg/kg infusion every two weeks. Subjects that experience a second virologic failure will be discontinued from the study. The total duration of study treatment will be 48 weeks, with the primary endpoint at Week 24.

ELIGIBILITY:
Inclusion Criteria:

Subjects must have all of the following to be included in the study:

* Triple-class experience, with no minimum exposure to any class (historical exposure to NRTI, NNRTI, PI)
* Cumulative HAART experience for a minimum of 6 months
* Virus susceptibility to one or more antiretroviral drugs in their selected OBT as determined by the PhenoSenseGT or similar assay and medication history
* Stable plasma HIV-1 RNA levels quantitated by reverse-transcriptase polymerase chain reaction (RT-PCR) of 10,000 copies/mL within 8 weeks prior to randomization (Day 1), while receiving a stable HAART regimen for a minimum of 4 weeks prior to screening. Stable viral load is defined as a difference of 0.5-log10 in HIV-1 RNA copies/mL from two measurements obtained at least 48 hours apart during the screening period
* Subjects must be failing their current HAART regimen or have discontinued a failing HAART regimen within 8 weeks prior to screening (screening visit 1)
* CD4+ cell count 50 cells/mL
* If sexually active, willingness to use an effective, medically accepted (including barrier) method of contraception during the study. To prevent superinfection, any male subject and the male sexual partner of any study subject should use a condom. All study subjects and all of their sexual partners should practice additional safe sex techniques to prevent spread of HIV.

Exclusion Criteria:

Subjects with any of the following characteristics will be excluded from the study:

* Any significant diseases (other than HIV infection) or clinically significant findings, including psychiatric and behavioral problems, medical history and/or physical examination, determined from screening, that, in the investigator's opinion, would preclude the subject from participating in this study
* Acute illness within one week prior to administration of study drug (including diarrhea and/or vomiting and fever and/or other signs and symptoms of infection such as leukocytosis, etc.)
* Any active infection secondary to HIV, requiring acute therapy. However, subjects that require maintenance therapy (i.e. secondary prophylaxis for opportunistic infections) will be eligible for the study
* Any immunomodulating therapy or systemic chemotherapy within 12 weeks prior to randomization (Day 1)
* Any investigational drug use within 30 days prior to randomization (Day 1). This does not include investigational drugs for the treatment of HIV-1 (NRTI, NNRTI or PI) under expanded access. OBT may include drugs not currently approved, but prescribed under expanded access (limited to NRTI's, NNRTI's and PI's).
* Any prior participation in an HIV vaccine study
* Opportunistic infections (OIs) in the previous 12 weeks prior to randomization (Day 1)
* Any prior exposure to TNX-355 (Hu5A8)
* Vaccination within 21 days (3 weeks) prior to randomization (Day 1)
* Any previous exposure to any virus/fusion entry inhibitor/s
* Any previous exposure to a monoclonal antibody (prior treatment with hepatitis B immune globulin [HBIG] or intravenous immune globulin [IVIG] is acceptable)
* Life expectancy of less than 12 months
* Female subjects who are either pregnant or breastfeeding
* Any illicit intravenous drugs within 6 months prior to randomization (Day 1)
* Any current alcohol or illicit drug use that, in the investigator's opinion, will interfere with the subject's ability to comply with the dosing schedule and protocol evaluations
* Clinically significant laboratory findings obtained during screening including:

  * Serum creatinine or BUN (>1.5 X Upper Limit of Normal [ULN])
  * Alkaline phosphatase, aspartase aminotransferase (AST), alanine aminotransferase (ALT) (any > 2.5 [ULN])
  * Total bilirubin (>1.5 ULN)
  * Pancreatic amylase and/or lipase (>1.5 ULN)
  * Hemoglobin (<9.0 g/dL for males; < 8.0 g/dL for females)
  * Platelet Count (<75,000 x 106/L)
  * Absolute Neutrophil Count (< 1,000 X 106/L)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2004-03

CONTACTS AND LOCATIONS:
Locations (15):
- United States (13):
  - Body Positive, Phoenix, Arizona
  - Altamed Corporation, Los Angeles, California
  - Tower ID Medical Associates, Los Angeles, California
  - Dupont Circle Physicians Group, Washington D.C., District of Columbia
  - IDC Research Initiative, Altamonte Springs, Florida
  - Bach and Godofsky, Bradenton, Florida
  - University of Miami, Miami, Florida
  - Comprehensive Research Institute, Tampa, Florida
  - Brobson Lutz, MD, LLC, New Orleans, Louisiana
  - Chase-Brexton Health Services, Inc., Baltimore, Maryland
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Tanox, Inc., Houston, Texas
- Sunnybrook Health Science Centre, Toronto, Ontario, Canada
- Clinical Research Puerto Rico, Inc., San Juan, Puerto Rico

REFERENCES:
- [Derived] Gathe JC, Hardwicke RL, Garcia F, Weinheimer S, Lewis ST, Cash RB. Efficacy, Pharmacokinetics, and Safety Over 48 Weeks With Ibalizumab-Based Therapy in Treatment-Experienced Adults Infected With HIV-1: A Phase 2a Study. J Acquir Immune Defic Syndr. 2021 Apr 1;86(4):482-489. doi: 10.1097/QAI.0000000000002591. PMID 33427765
- See also: Tanox, Inc. website — http://www.tanox.com